CLINICAL TRIAL: NCT05597111
Title: Comparison of Docosahexaenoic Acid (DHA) Serum and Cervical Mucus Sample Values in Patients With Polycystic Ovary Syndrome (PCOS) and Control Group
Brief Title: Comparison of Docosahexaenoic (DHA) Values in Patients With Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Kagitci, Assistant professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2022/183
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Docosahexaenoic acid; inflammation; omega-3
MeSH Terms: conditions — Polycystic Ovary Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Blood DHA levels of patients with PCOS: The patients diagnosed as PCOS according to Rotterdam criteria will be the study group. The DHA leves in blood sample of the patients will be recorded
  Interventions: Diagnostic Test: DHA levels of blood and cervical mucus
- BloodDHA levels of the control group: The patients without PCOS will be control group. The DHA leves in blood sample of the patients will be recorded
  Interventions: Diagnostic Test: DHA levels of blood and cervical mucus

INTERVENTIONS:
Diagnostic Test: DHA levels of blood and cervical mucus — DHA levels of blood and cervical mucus of the control and the study groups will be measure

SUMMARY:
Although PCOS has been known for many years, its etiology and treatment are not clearly known. The prevalence of PCOS varies between populations. It is a familial endocrinolpathology with a chronic course, multifactorial, polygenic feature seen with an average prevalence of 6-8% in women in the reproductive period.Chronic inflammation is involved in the pathophysiology of many chronic diseases. PCOS, which is a proinflammatory condition, has been associated with insulin resistance and hyperandrogenism in previous studies.

Omega-3 fatty acids have anti-inflammatory, anti-thrombotic, anti-arrhythmic properties, reducing lipid levels such as serum triglyceride and LDL cholesterol, and having positive effects on the immune system. Therefore, their deficiencies include fatigue, joint pain, frequent infections, etc. is seen. Omega-6 fatty acids have the opposite effect.

DHA is a member of the omega-3 fatty acids family. Dietary components play an important role in chronic inflammation.

According to our literature review, there is no study that detects docosahexaenoic acid (DHA) levels in blood and cervical mucus samples in patients with PCOS. We think that we will contribute to the diagnosis and treatment processes of PCOS patients by detecting DHA levels in this study.

In this study, we aim to compare the values of docosahexaenoic acid (DHA) in serum and cervical mucus samples in patients with polycystic ovary syndrome with the control group.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) was first described in 1935 by Dr. Stein and Dr. It was defined by Leventhal. Although PCOS has been known for many years, its etiology and treatment are not clearly known. The prevalence of PCOS varies between populations. It is a familial endocrinolpathology with a chronic course, multifactorial, and polygenic features, with an average prevalence of 6-8% in women in the reproductive period. PCOS is a symptom complex that requires a multidisciplinary approach involving many departments. The clinic in PCOS progresses with different symptoms in each patient. In general, such as menstrual irregularities, alopecia due to androgen excess, acne, hirsutism, infertility, obesity, abnormal lipid levels, glucose intolerance, acanthosis nigricans, Type 2 diabetes, endometrial hyperplasia, endometrial cancer, ovarian cancer, breast cancer, hypertension, coronary heart diseases. It progresses with mood changes ,cardiovascular diseases, abortion, IUGR, depression, anxiety, eating disorders, and obstructive sleep apnea. Determining the diagnostic criteria for PCOS is important in terms of long-term risks rather than short-term effects in patients. PCOS diagnostic criteria were divided into different categories in 3 different periods. For the first time, 3 important criteria were determined in the National Institutes of Health Criteria (NICHD) in 1990. (1)menstrual dysfunction (oligo/anovulation), (2) hyperandrogenism/hyperandrogenemia (hirsutism, acne, androgenetic alopecia), (3) causes mimicking similar clinics should be excluded. Rotterdam Consensus Criteria was determined in 2003 for the second time in the diagnosis of PCOS. Rotterdam Criteria At least 2 of the 3 major criteria must be present. The first criterion is (1) menstrual dysfunction (oligo/anovulation), (2) hyperandrogenism/hyperandrogenemia (hirsutism, acne, androgenetic alopecia), (3) polycystic ovarian morphology in ultrasonography (at least one ovary with 12 or more follicles 2-9 mm in diameter) and ovarian volume of 10 ml or more) and similar clinical mimicking causes should be excluded. Third are the Androgen Excess Society (AE-PCOS) criteria made in 2006. The criteria should be (1) menstrual dysfunction (oligo/anovulation), (2) hyperandrogenism/hyperandrogenemia (hirsutism, acne, androgenetic alopecia), (3) polycystic ovary appearance on ultrasonography, and (a) causes mimicking similar clinics. 1 and 2 or 2 and 3 conditions were determined from these criteria.

Chronic inflammation is involved in the pathophysiology of many chronic diseases. PCOS, which is a proinflammatory condition, has been associated with insulin resistance and hyperandrogenism in previous studies.

All fats play important roles in energy metabolism and body functions; however, the omega-6 precursor, linoleic acid (LA), and the omega-3 precursor, alpha-linolenic acid (ALA), are known as essential fatty acids because they cannot be synthesized in the body and therefore become a vital component of a healthy diet. These are unsaturated fatty acids with double bonds between carbon atoms, unlike saturated fatty acids, where all carbon atoms are "saturated" with hydrogen atoms. Depending on the position of the double bond with respect to the methyl end carbon (omega carbon), unsaturated fatty acids are classified as omega-3 and omega-6 fatty acids. Omega-3 fatty acids such as eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) contain alpha- it is derived from linolenic acid (ALA) .

Omega-3 fatty acids have anti-inflammatory, anti-thrombotic, anti-arrhythmic properties, reducing lipid levels such as serum triglyceride and LDL cholesterol, and having positive effects on the immune system. Therefore, their deficiencies include fatigue, joint pain, frequent infections, etc. is seen. Omega-6 fatty acids have the opposite effect.

DHA is a member of the omega-3 fatty acids family. Dietary components play an important role in chronic inflammation. It has been reported that a diet rich in omega-3 fatty acids may have positive effects on epigenomes. It has been shown that inflammatory cytokines such as interleukin 1-β, thromboxane A2, interleukin-6, tumor necrosis factor, leukotriene B and C-reactive protein increase in chronic diseases. In particular, the anti-inflammatory effects of omega-3 fatty acids such as eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) have been reported.

There are studies showing that some inflammatory substances in the endometrial washings of PCOS patients are different from the normal population . These studies suggest that inflammation may also be a cause of common infertility in PCOS patients by affecting endometrial receptivity.

According to our literature review, there is no study that detects docosahexaenoic acid (DHA) levels in blood and cervical mucus samples in patients with PCOS. We think that we will contribute to the diagnosis and treatment processes of PCOS patients by detecting DHA levels in this study.

In this study, we aim to compare the values of docosahexaenoic acid (DHA) in serum and cervical mucus samples in patients with polycystic ovary syndrome with the control group.

ELIGIBILITY:
Inclusion Criteria:

1- Patients with polycystic ovary syndrome

Exclusion Criteria:

1. Pregnancy
2. Malignity
3. postmenopause
4. diagnosis of congenital adrenal syndrome
5. Oral contraseptive use at last 3 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: the patients diagnosed as PCOS according to Rotterdam criteria will be accepted as study group
Sampling Method: Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Blood DHA levels of patients with PCOS | 3 months
  Blood DHA levels of patients with PCOS
Cervical mucus DHA levels of patients with PCOS | 3 months
  Cervical mucus DHA levels of patients with PCOS

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan Univercity, Rize, Turkey (Türkiye)